CLINICAL TRIAL: NCT01343121
Title: Measurement of Gemcitabine Metabolites in Blood and Urine as Predictors of Response to GemX Bladder Radiotherapy
Acronym: Gemtrans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10_DOG04_124
Record Dates: First submitted 2011-04-07; First posted 2011-04-27 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Bladder Cancer
Keywords: Radiotherapy; GemX Chemoradiotherapy; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sample collection (Other): This is a single arm study. Patients will be seen on day 1, 8, 15 and 22 and will have the following samples collected:
  * Pre gemcitabine urine sample
  * Blood sample 30 minutes post Gemcitabine infusion
  * Urine and blood sample 2 hours post Gemcitabine infusion
  Interventions: Other: sample collection

INTERVENTIONS:
Other: sample collection — Blood samples will be collected on days 1, 8, 15 and 22. They will be taken 30 minutes and 2 hours post Gemcitabine infusion.
Other: sample collection — Urine will be collected on days 1, 8, 15 and 22. They will be taken pre gemcitabine and 2 hours post Gemcitabine
Other: Sample Collection — Quality of Life (QOL) questionnaires given to the patient at each visit

SUMMARY:
The purpose of this study is to test the hypothesis that plasma, peripheral blood mononuclear cell and urine levels of Gemcitabine and its metabolites, 30 mins or 2 hours post infusion, predict response to GemX chemoradiation at first check cystoscopy, 3 months from the end of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of muscle-invasive transitional cell carcinoma.
* suitable for treatment with radical concurrent chemoradiotherapy with GemX.
* Standard radiological assessments with CT or MR for staging.
* ECOG performance status 0-2
* Adequate pre-treatment haematological and biochemical parameters
* Age greater than or equal to 18 years
* No significant co-morbidity thereby excluding patient from having radical treatment.
* No previous treatment for diagnosis of muscle-invasive bladder cancer or other pelvic radiotherapy.
* Women of child bearing age MUST have a negative pregnancy test prior to study entry and be using an adequate contraception method, which must be continued for 3 months after the study, unless child bearing potential has been terminated by surgery/radical radiotherapy
* Patients must have given written informed consent

Exclusion Criteria:

* Patients with a known history of anaphylactic reaction to any other drug.
* Patients must not have a history of other malignant diseases other than adequately treated non-melanotic skin cancer or in-situ carcinoma of the uterine cervix
* Any evidence of severe or uncontrolled systemic diseases which, in the view of the investigator, makes it undesirable for the patient to participate in the trial.
* Evidence of significant clinical disorder or laboratory finding which, in the opinion of the investigator makes it undesirable for the patient to participate in the trial Any other serious uncontrolled medical conditions
* Clinical evidence of metastatic disease to brain
* Any pregnant or lactating woman
* Any patient with a medical or psychiatric condition that impairs their ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02-02 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2017-11-24 (Actual)

PRIMARY OUTCOMES:
Does response at Cystoscopy correlate with results of sample analysis | 3 months following the end of GemX chemoradiation
  To test the hypothesis that plasma, peripheral blood mononuclear cell and urine levels of gemcitabine and its metabolites, 30 mins or 2 hrs post-infusion, predict response to GemX chemoradiation at first check cystoscopy, 3 months from the end of radiotherapy. Gemcitabine will be measured in plasma by HPLC-MS using a published validated method. We have developed an assay for intracellular gemcitabine triphosphate which should determine levels in PBMCs from 10 - 15 ml blood. Response at Cystoscopy is measured as either complete response, superficial disease or muscle-invasive disease.

SECONDARY OUTCOMES:
cause-specific and overall survival rates | 3 years
acute and late toxicities as assessed by RTOG and LENT SOM scales | 3 years
  Toxicity is measured using LENT-SOMA (patient-reported) and CTCAE v4.0 (clinical assessment) during treatment and at follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Ananya Choudhury, Phd, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, Gtr Manchester, United Kingdom